CLINICAL TRIAL: NCT01591031
Title: Laryngeal Injuries After Anesthesia Induction With Sevoflurane and After Anesthesia Induction With Rocuronium. A Randomized, Prospective, Controlled Trial
Brief Title: Laryngeal Injuries After Anesthesia Induction With Sevoflurane and After Anesthesia Induction With Rocuronium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Thomas Mencke, Principal Invastigator, Clinical Associate Professor, Dr. Thomas Mencke, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A 2011 124
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Laryngeal Injuries
Keywords: laryngeal injuries; vocal cord injuries; hoarseness; sore throat
MeSH Terms: conditions — Hoarseness; Pharyngitis | interventions — Sevoflurane; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevoflurane (Active Comparator): anesthesia induction with propofol, remifentanil and sevoflurane
  Interventions: Drug: Sevoflurane
- rocuronium (Active Comparator): anesthesia induction with propofol, remifentanil and rocuronium
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Sevoflurane — anesthesia induction with propofol, remifentanil and sevoflurane; afterwards tracheal intubation
  Arms: sevoflurane
Drug: Rocuronium — anesthesia induction with propofol, remifentanil and rocuronium; afterwards tracheal intubation
  Arms: rocuronium

SUMMARY:
Anesthesia induction with sevoflurane is not associated with an increased incidence or severity of laryngeal injuries compared with an anesthesia induction with a muscle relaxant.

ELIGIBILITY:
Inclusion Criteria:

* ear-nose-throat surgery
* orotracheal intubation for surgery of the ear

Exclusion Criteria:

* obesity
* allergy against the study drugs
* patients with a known or suspected difficult airway (Mallampati score 3 or 4 and a mouth opening < 3.5 cm).
* all patients were examined by stroboscopy one day before surgery and were excluded from the study when preexisting pathologies of the vocal cords were found

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
incidence of vocal cord injuries | 24 h after tracheal intubation

SECONDARY OUTCOMES:
incidence of hoarseness | 24h, 48 h, and 72 h after tracheal intubation
incidence of soar throat | 24h, 48h, and 72 h after tracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Mencke T, Jacobs RM, Machmueller S, Sauer M, Heidecke C, Kallert A, Pau HW, Noeldge-Schomburg G, Ovari A. Intubating conditions and side effects of propofol, remifentanil and sevoflurane compared with propofol, remifentanil and rocuronium: a randomised, prospective, clinical trial. BMC Anesthesiol. 2014 May 22;14:39. doi: 10.1186/1471-2253-14-39. eCollection 2014. PMID 24860256